CLINICAL TRIAL: NCT02816632
Title: Feedbacks' Influence on Decision Making Processes
Acronym: Feedbacks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL15_0221; 2015-A00623-46 (Other: ID-RCB)
Record Dates: First submitted 2016-06-20; First posted 2016-06-28 (Estimated); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers
Keywords: functional Magnetic Resonance Imaging; Galvanic Vestibular Stimulation; Feedback Processing; Reward, Social, Vestibular System; Cingulate Cortex; Decision-making

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- healthy volunteers (Experimental)
  Interventions: Other: mRI; Other: Effect of Galvanic Vestibular Stimulation on decision making processes

INTERVENTIONS:
Other: mRI — Neural bases of feedbacks' influence on decision making processes
Other: Effect of Galvanic Vestibular Stimulation on decision making processes — Galvanic Vestibular Stimulation (GVS) stimulates the vestibular system through low intensity electric currents applied at the basis of the VIII cranial nerve, upon the mastoid processes. In the Right-Anodal condition the positive electric charge is applied through electrodes placed upon the right mastoid and it mainly activates structures within the left brain hemisphere. In the Left-Anodal condition the positive electric charge is applied through electrodes placed upon the left mastoid and it mainly activates structures within the right brain hemisphere. In the SHAM condition, low intensity electric currents are applied 5 cm below the mastoid processes. This condition does not activate the vestibular system and serves as a control condition to account for unspecific activating effects of all electric stimulations (e.g., arousal, discomfort). The three conditions will be applied in three different sessions (i.e. days) in randomized order.

SUMMARY:
The purpose of this research is to identify and probe the neural networks involved in feedback processing. It aims at translating this knowledge to clinical populations in which this network is disrupted or compromised.

It includes two studies: 1) with fMRI in healthy subjects to identify the neural bases of feedback processing on decision making using different types of feedback (neutral, social and monetary) presented either infra- or supra-laminary and 2) probing the role of one structure, the anterior cingulate cortex, using Galvanic Vestibular Stimulation (GVS) in healthy subjects. The interventional part consists in the administration of Galvanic Vestibular Stimulation (GVS), which by means of small intensity currents activates the vestibular organs and subsequently vestibular-related brain areas. GVS will be delivered to healthy participants engaged in behavioural tasks requiring the processing of feedbacks of different nature (e.g. social or monetary feedbacks)

ELIGIBILITY:
Inclusion Criteria:

* Benefit of social health security
* Normal or corrected-to-normal vision

Exclusion Criteria:

* Anamnesis of neurological of psychiatric illness
* Pregnancy or breastfeeding
* Administrative measures restricting legal rights
* Epilepsy (including familiarity), migraines, chronic headaches
* presence of pacemakers, cochlear implants, surgical clips, or any metallic component fixed in participants' body
* Current treatment with psychotropic drugs
* Alcohol assumption during the last 24 hours
* Sleep deprivation
* Recent participation to other brain stimulation studies (< 1 week)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

PRIMARY OUTCOMES:
Behavioral performance (Accuracy) | up to 4 days
  The proportion of correct responses, automatically computed by professional programs (e.g. Presentation) running on standard Personal Computers depending on different contexts (e.g. different feedback: neutral, social and monetary).
Behavioral performance (Reaction times) | up to 4 days
  The proportion of reaction times provided, automatically computed by professional programs (e.g. Presentation) running on standard Personal Computers depending on different contexts (e.g. different feedback: neutral, social and monetary).

SECONDARY OUTCOMES:
Neural activity (BOLD signal measured using fMRI) as a function of the nature of the feedback. | up to 4 days
  Neural activity changes during learning of visuomotor associations in different contexts (e.g. different feedback: neutral, social and monetary) measured using Blood-oxygen-level dependent contrast imaging (BOLD).

CONTACTS AND LOCATIONS:
Overall Officials: Caroline TILIKETE, MD, Principal Investigator — Unité de Neuro-Ophtalmologie Hôpital Neurologique - HOSPICES CIVILS DE LYON
Locations (1):
- Unité de Neuro-Ophtalmologie Hôpital Neurologique - HOSPICES CIVILS DE LYON, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blini E, Tilikete C, Farne A, Hadj-Bouziane F. Probing the role of the vestibular system in motivation and reward-based attention. Cortex. 2018 Jun;103:82-99. doi: 10.1016/j.cortex.2018.02.009. Epub 2018 Feb 27. PMID 29574253
- [Background] Blini E, Tilikete C, Chelazzi L, Farne A, Hadj-Bouziane F. The role of the vestibular system in value attribution to positive and negative reinforcers. Cortex. 2020 Dec;133:215-235. doi: 10.1016/j.cortex.2020.09.004. Epub 2020 Oct 2. PMID 33130427